CLINICAL TRIAL: NCT06521853
Title: Comparison Between PEEK With Autogenous Bone Graft and PEEK With Xenograft in Maxillary Sinus Augmentation: Clinical, Radiographic and Histomorphometric Analysis. Randomized Clinical Trials.
Brief Title: Comparison Between PEEK With Autogenous Bone Graft and PEEK With Xenograft in Maxillary Sinus Augmentation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, mohamed gamal hammad, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 33-6-23
Record Dates: First submitted 2024-04-17; First posted 2024-07-26 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Maxillary Sinus
Keywords: maxillary sinus augmentation ; bone graft
MeSH Terms: interventions — polyetheretherketone; Transplantation, Heterologous

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PEEK With Autogenous Bone Graft (Experimental): maxillary sinus elevation using PEEK device and placement of autogenous bone graft
  Interventions: Other: PEEK With Autogenous Bone Graft
- PEEK With Xenograft (Experimental): maxillary sinus elevation using PEEK device and placement of xenograft
  Interventions: Other: PEEK With Xenograft

INTERVENTIONS:
Other: PEEK With Autogenous Bone Graft — placement of PEEK With Autogenous Bone Graft
  Arms: PEEK With Autogenous Bone Graft
Other: PEEK With Xenograft — placement of PEEK With xenograft
  Arms: PEEK With Xenograft

SUMMARY:
Comparison Between PEEK With Autogenous Bone Graft and PEEK With Xenograft in Maxillary Sinus Augmentation

DETAILED DESCRIPTION:
Comparison Between PEEK With Autogenous Bone Graft and PEEK With Xenograft in Maxillary Sinus Augmentation: clinical, radiographic and histomorphometric analysis .

ELIGIBILITY:
Inclusion Criteria:

* posterior edentulous ridge less than 4mm in bone height

Exclusion Criteria:

* insufficient oral hygiene and motivation

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
bone height | after 6 months
  using CBCT in mm

SECONDARY OUTCOMES:
bone quality | after 6 months
  core biopsy (Histomorphometric evaluation)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of dentistry Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No